CLINICAL TRIAL: NCT03727438
Title: Provider Supported Self-Help Cognitive Behavioral Therapy for Insomnia (Tele-Self-CBTI)
Brief Title: Tele-Self CBTI Trial
Acronym: Tele-Self CBTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 16-281; 1I01HX002350-01A2 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Insomnia Disorder
Keywords: Cognitive Behavioral Therapy for Insomnia; Self-Directed Treatment; Telehealth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-Self CBTI (Experimental): Tele-Self CBTi is a telephone-based CBT insomnia intervention
  Interventions: Behavioral: Tele-Self CBTI
- Health Education Control (Active Comparator): The Health Education is an active control arm
  Interventions: Other: Health Education Control

INTERVENTIONS:
Behavioral: Tele-Self CBTI — The Tele-Self CBTI intervention is comprised of two treatment components: 1) self-directed treatment via weekly readings from a treatment manual, and 2) weekly telephone-based nurse support contacts across a 8 week intervention period. Participants have 8 weeks to complete 6 study-related phone calls
  Arms: Tele-Self CBTI
Other: Health Education Control — The Health Education Control condition is comprised of two components: 1) weekly reading from a health education manual, and 2) weekly telephone-based nurse support contacts across a 8 week period. At the end of the study, participants in the Health Education arm will be offered assistance for their sleep complaints, as needed, through the Durham Behavioral Sleep Medicine clinic.
  Other Names: Control
  Arms: Health Education Control

SUMMARY:
Insomnia is one of the most common complaints among service-members and Veterans of recent military conflicts. Insomnia has been shown to play a causal role in mental health, hypertension, obesity, and other health conditions, increasing risk for all-cause mortality. Cognitive-Behavioral Therapy for Insomnia (CBTI) produces both short-term and sustained resolution of insomnia with fewer adverse side effects than medications, but access to behavioral sleep medicine expertise within the VA is very limited.

This study compares Tele-Self CBTI to Health Education Control for improved insomnia severity among treatment-seeking Veterans with Insomnia. In this study, 200 participants will be randomized with a 50/50 chance to either Tele-Self CBTI or a Health Education Control condition. Eligible participants are Veterans who are: a) prescribed sleep medications; b) diagnosed with insomnia; and/or c) referred for clinic-based CBTI (but not yet treated) for insomnia. Participants will be identified using electronic health records (EHR) and telephone interviews.

Participants' sleep will be assessed at three time points, at Baseline, 8 weeks and 6 months after Baseline. The Tele-Self CBTi intervention is comprised of two treatment components: 1) self-directed treatment via weekly readings from a treatment manual, and 2) weekly telephone-based nurse support contacts across a 8 week intervention period. Participants randomized to Tele-Self CBTI will complete 6 weekly readings in addition to having 6 weekly telephone contacts with a study nurse; each call lasting approximately 20 minutes. Patients randomized to Health Education Control (HEC) will receive a health education manual on 6 health topics. They will also complete 6 weekly readings from the HEC manual and receive 6 weekly telephone contacts from a study nurse. All participants will continue to receive usual medical care while participating in the study. Following completion of this 6 month study, participants randomized to HEC and interested in additional help for their sleep will be referred to the Durham VA Behavioral Sleep Medicine Clinic.

DETAILED DESCRIPTION:
Insomnia is one of the most common complaints among service-members and Veterans of recent military conflicts. Insomnia diagnoses increased 19-fold among military service members from 2000 to 2009. Insomnia has been shown to play a causal role in depression, anxiety, suicidality, disability due to a mental health disorder, hypertension, obesity, metabolic syndrome, diabetes, and all-cause mortality, thus serving as an additional risk factor for some of the most common medical conditions seen in patients utilizing the VA healthcare system. Cognitive-Behavioral Therapy for Insomnia (CBTI) produces both short-term and sustained resolution of insomnia with fewer adverse side effects than pharmacotherapy. But access to behavioral sleep medicine expertise within the VA is very limited.

Self-management and telehealth are viable options for achieving these goals. This study is a randomized controlled trial comparing Tele-Self CBTI to Health Education Control (HEC) for improved insomnia severity among treatment-seeking Veterans with Insomnia. In this 2-arm trial, 200 participants will be randomized in a 1:1 ratio to Tele-Self CBTI or a Health Education Control condition. Eligible participants are Veterans who are: a) prescribed sleep medications; b) diagnosed with insomnia; or c) referred for clinic-based CBTI (but not yet treated) will be identified using electronic health records (EHR) and telephone interviews.

Outcomes include insomnia severity in addition to subjective (sleep diary) and objective (actigraphy) measures of sleep variables, including: sleep onset latency (SOL), wakefulness after sleep onset (WASO), and sleep efficiency (SE). These outcomes will be assessed at 3 time points: baseline, 8 weeks, and 6 months after baseline. Participants in both arms will continue to receive usual medical care. Each assessment period involves: a) 2 weeks of home-based sleep assessment (diary and actigraphy), and b) completion of telephone-based questionnaires. Following completion of each home-based sleep assessment period, a study staff member will contact participants to complete study questionnaires by phone. Study participants will be asked to return actigraphy devices at the end of each assessment period.

Tele-Self CBTI is comprised of two treatment components: 1) Self-directed treatment via a treatment manual entitled, "Improve your Sleep: A Self-Guided Approach for Veterans with Insomnia" and 2) telephone-based nurse support. Participants will complete 6 weekly reading modules from the treatment manual on topics reflecting typical CBTI treatment components: Sleep Restriction; Stimulus Control; Cognitive Therapy; Relaxation; and Sleep Hygiene Education. Tele-Self CBTI will be delivered across 6 weekly telephone contacts of 20 minutes or less through a study nurse who will briefly review treatment manual content with the participant, review sleep diaries, and create and adjust sleep prescriptions as needed. Patients randomized to Health Education Control (HEC) will completed weekly readings and receive 6 weekly phone calls from a study nurse. Consistent with phone contacts in the intervention arm, HEC phone contacts will involve reviewing content in the health education manual and will last approximately 20 minutes; matching as closely as possible call duration with Tele-Self CBTI participants. Sleep-focused content will be prohibited during HEC calls. Participants have 8 weeks to complete the 6 phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for Insomnia Disorder
* Receives care through the Durham VA Health Care System (HCS) catchment area

Exclusion Criteria:

* Severe Obstructive Sleep Apnea with treatment non-adherence
* Unstable co-morbid sleep disorder determined via chart review

  * e.g., rule out for Narcolepsy, rule out for Shift Work Disorder
* Current or prior participation in Cognitive Behavioral Therapy for Insomnia (CBTI)
* Excessive daytime sleepiness
* Nighttime or rotating shift work within the last year
* Psychotic disorder diagnosis
* Bipolar disorder diagnosis
* Recreational substance use
* Current alcohol abuse
* Severe depression or suicidality
* Dementia diagnosis
* Cognitive impairment
* Epilepsy diagnosis
* Seizure disorder diagnosis
* Lack of proficiency in the English language
* Hearing impairment that impedes telehealth intervention
* Unable to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christi S. Ulmer, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulmer CS, McCant F, Stechuchak KM, Olsen M, Bosworth HB. Prevalence of insomnia disorder and sleep apnea in a sample of veterans at risk for cardiovascular disease. J Clin Sleep Med. 2021 Jul 1;17(7):1441-1446. doi: 10.5664/jcsm.9228. PMID 33688827
- [Result] Ulmer CS, Bosworth HB, Zervakis J, Goodwin K, Gentry P, Rose C, Jeffreys AS, Olsen MK, Weidenbacher HJ, Beckham JC, Voils CI. Provider-supported self-management cognitive behavioral therapy for insomnia (Tele-Self CBTi): Protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Feb;125:107060. doi: 10.1016/j.cct.2022.107060. Epub 2022 Dec 22. PMID 36567058
- [Result] Ulmer CS, Voils CI, Jeffreys AS, Olsen M, Zervakis J, Goodwin K, Gentry P, Rose C, Weidenbacher HJ, Beckham JC, Bosworth HB. Nurse-Supported Self-Directed Cognitive Behavioral Therapy for Insomnia: A Randomized Clinical Trial. JAMA Intern Med. 2024 Nov 1;184(11):1356-1364. doi: 10.1001/jamainternmed.2024.4419. PMID 39250131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were veterans recruited from the Durham VA Health Care System (HCS) catchment area between 10/4/2019 to 4/26/2022. A data pull from the electronic medical record (EMR), identified veterans who were seeking treatment for insomnia but not yet treated using CBT-I. A chart review of the electronic record was also performed. Potentially eligible patients were then mailed an invitation letter beginning on 9/20/19. They were then contacted, consented and screened over the phone.
Pre-assignment Details: Consented participants completed a 2 week assessment period before being randomized. Participants not completing at least 10 days of sleep diary and/or baseline questionnaires were excluded, even if they provided actigraphy data. 178 completed baseline, enrolled and randomized to either Tele-Self CBTI or Health Education Control (HEC), using a stratified, blocked randomization, by baseline Insomnia Severity Index score (≤20/>20) and presence/absence of a pre-existing mental health diagnosis.
Groups:
- Tele-Self CBTI: The Tele-Self CBTI intervention is comprised of two treatment components: 1) self-directed treatment via weekly readings from a treatment manual, and 2) weekly telephone-based nurse support contacts across a 8 week intervention period.
Period: Baseline
Arm/Group | Tele-Self CBTI | Health Education Control
Started | 88 | 90
Completed | 88 | 90
Not Completed | 0 | 0
Period: Intervention Period
Arm/Group | Tele-Self CBTI | Health Education Control
Started | 88 | 90
Completed | 77 | 88
Not Completed | 11 | 2
Not completed — Did not complete at least 3 calls but remained in study | 7 | 1
Not completed — Excluded (health) | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Period: 8 Week Assessment
Arm/Group | Tele-Self CBTI | Health Education Control
Started | 84 (Participants who did not complete the 8 week assessment due to being unable to be reached or protocol deviation were not excluded from the study. Lost to follow-up status was determined at the 6 month assessment period.) | 89 (Participants who did not complete the 8 week assessment due to being unable to be reached or protocol deviation were not excluded from the study. Lost to follow-up status was determined at the 6 month assessment period.)
Completed | 70 (Due to study error 2 participants were not contacted to begin study procedures during the 8 week assessment window.) | 83
Not Completed | 14 | 6
Not completed — Did not complete assessment but remained in study | 6 | 5
Not completed — Did not complete due to study error, remained in study | 2 | 0
Not completed — Withdrawal by Subject | 6 | 1
Period: 6 mo Assessment
Arm/Group | Tele-Self CBTI | Health Education Control
Started | 78 | 88
Completed | 68 (10 CBTI withdrawals consists of: 3 during intervention period, 1 after intervention but before 8 week, 2 at 8 week and 4 at 6 months) | 77 (1 additional participant did not complete 2 items on the ISI and was not included in the 6 mo analysis (n=76). 7 HEC withdrawals consists of: 1 during intervention period, 1 at 8 week, and 5 at 6 month.)
Not Completed | 10 | 11
Not completed — did not complete assessment | 10 | 11

BASELINE CHARACTERISTICS:
Population: Overall number stratified by intervention. Does not include participants consented but not randomized.
Groups:
- Tele-Self CBTI: The Tele-Self CBTI intervention is comprised of two treatment components: 1) self-directed treatment via weekly readings from a treatment manual, and 2) weekly telephone-based nurse support contacts across a 6 week intervention period.
- Health Education Control: The Health Education Control condition is comprised of two components: 1) weekly reading from a health education manual, and 2) weekly telephone-based nurse support contacts across a 6 week period. At the end of the study, participants in the Health Education arm will be offered assistance for their sleep complaints, as needed, through the Durham Behavioral Sleep Medicine clinic.
- Total: Total of all reporting groups
Arm/Group | Tele-Self CBTI | Health Education Control | Total
Number analyzed (Participants) | 88 | 90 | 178
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 55.1 (13.2) | 55.1 (13.3) | 55.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 62 | 66 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 81 | 86 | 167
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 42 | 76
  White | 47 | 40 | 87
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 90 | 178
Baseline ISI >20 n (%) [Count of Participants; unit: Participants] — Having a baseline Insomnia Severity Index (ISI) is 20 or greater (count)
  Participants | 17 | 18 | 35
Mental health diagnosis n (%) [Count of Participants; unit: Participants] — participant has one (or more) mental health diagnosis listed in medical record
  Participants | 73 | 74 | 147
Currently using sleep medications n [Count of Participants; unit: Participants] | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity
Description: Insomnia Severity Index (ISI): The ISI is recommended as the standard for self-reported insomnia symptoms, and will be used as the primary outcome measure. The ISI is a 7-item questionnaire providing a global measure of perceived insomnia severity. Each item is rated on a 5-point Likert scale and the total score ranges from 0 (no reported symptoms) to 28 (highest insomnia severity symptoms). The following guidelines are recommended for interpreting the total score: 0-7 (no clinical insomnia), 8-14 (sub threshold insomnia), 15-21 (insomnia of moderate severity), and 22-28 (severe insomnia). In clinical samples, a cut off score of 11 was shown to have the greatest sensitivity and specificity for correctly identifying study participants meeting criteria for insomnia diagnosis.
Time Frame: Baseline to 8 weeks
Population: This is an intention to treat analysis. All subjects who completed baseline were included in analysis. Estimated means were calculated from a linear mixed model and used for the analysis.
Measure: Mean (Standard Error); unit: ISI score
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 88 | 90
ISI score
  Baseline | 16.1 (0.2) | 16.1 (0.2)
  8 Weeks: number analyzed (Participants) | 70 | 83
  8 Weeks | 10.4 (0.5) | 14.1 (0.5)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Analyses were conducted according to the intention-to-treat principle. All available data, including observations from participants who dropped out of the study, were used for primary and secondary analyses. Our modeling estimation approach was conducted with full-likelihood methods, providing unbiased treatment effect estimates under a missing-data framework known as "missing at random" (MAR); Test type: Equivalence — alpha = .05; p < 0.01, Mixed Models Analysis — alpha=.05; Model parameters included a common intercept (baseline means constrained to be equal), stratification variables, timepoint, and arm by timepoint; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-5.0 to -2.4]

2. Secondary Outcome: Subjective Sleep Onset Latency (SOL)
Description: Sleep Diary sleep onset latency, using the Consensus Sleep Diary (CSD), which is the amount of time asleep in bed divided by the amount of time in bed, averaged across days. The investigators will use a call-in interactive Voice Response (IVR) approach to collect sleep diary data during each of the three 2-week assessment periods. Diary data will then be averaged across each 2-week assessment period.
Time Frame: Baseline to 8 week
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 88 | 90
minutes
  Baseline | 49.4 (2.6) | 49.4 (2.6)
  8 week: number analyzed (Participants) | 70 | 83
  8 week | 26.5 (3.1) | 46.1 (2.9)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Test type: Equivalence — alpha= .05; p < 0.01, Mixed Models Analysis — alpha = 0.05; Mean Difference (Final Values) = -19.6, 95% CI 2-sided [-26.7 to -12.5]

3. Secondary Outcome: Subjective Wake After Sleep Onset (WASO)
Description: Sleep Diary WASO, using the Consensus Sleep Diary (CSD). The investigators will use a call-in interactive Voice Response (IVR) approach to collect sleep diary data during each of the three 2-week assessment periods. Diary data will then be averaged across each 2-week assessment period to determine SOL, WASO and SE.
Time Frame: Baseline to 8 week
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 88 | 90
minutes
  Baseline | 58.8 (3.1) | 58.8 (3.1)
  8 week: number analyzed (Participants) | 70 | 83
  8 week | 33.5 (3.6) | 54.0 (3.3)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Test type: Equivalence — alpha = .05; p < 0.01, Mixed Models Analysis — alpha = .05; Mean Difference (Final Values) = -20.6, 95% CI 2-sided [-29.1 to -12.0]

4. Secondary Outcome: Subjective Sleep Efficiency (SE)
Description: Sleep Diary sleep efficiency, calculated from the Consensus Sleep Diary (CSD), which is the percent of the time asleep out of amount of time spent in bed. The investigators will use a call-in interactive Voice Response (IVR) approach to collect sleep diary data during each of the three 2-week assessment periods. Diary data are averaged across each 2-week assessment period.
Time Frame: Baseline to 8 week
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of time in bed where asleep
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 88 | 90
percentage of time in bed where asleep
  Baseline | 65.4 (1.2) | 65.4 (1.2)
  8 week: number analyzed (Participants) | 70 | 83
  8 week | 79.0 (1.5) | 68.0 (1.4)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Test type: Equivalence — alpha = .05; p < 0.01, Mixed Models Analysis; alpha = 0.05; Mean Difference (Final Values) = 11.0, 95% CI 2-sided [7.7 to 14.3]

5. Secondary Outcome: Objective Wake After Sleep Onset
Description: Objective WASO using Wrist Actigraphy: The investigators will use Actiwatch (Respironics, Inc.) wristwatch style actigraphs for collecting objective sleep data. Actiwatches contain a calibrated accelerometer that samples, digitizes, and stores movement activity. When interfaced with a computer, a scoring algorithm provides estimates of various sleep parameters. WASO is the total number of epochs between the start time and the end time of the given sleep interval scored as wake by Actiware software multiplied by the epoch length in minutes. The investigators will average data across each two-week assessment period. Not all participants completed actigraphy procedures
Time Frame: Baseline to 8 week
Population: To be included in actigraphy analyses, actigraphy data must have overlapped with sleep diary data (same dates) for a minimum of 7 nights. Estimated means were used. All available data, including observations from participants who dropped out of the study, were used for primary and secondary analyses. Model parameters included a common intercept (baseline means constrained to be equal), with the model examining estimated group differences.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 74 | 74
minutes
  Baseline | 48.7 (1.8) | 48.7 (1.8)
  8 week: number analyzed (Participants) | 54 | 63
  8 week | 48.7 (2.7) | 54.9 (2.6)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Test type: Equivalence — Alpha = .05; p > 0.05, Mixed Models Analysis — Alpha = .05; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-12.5 to 0.1]

6. Secondary Outcome: Objective Total Sleep Time (TST)
Description: Objective total sleep time using Wrist Actigraphy: The investigators will use Actiwatch (Respironics, Inc.) wristwatch style actigraphs for collecting objective sleep data. Actiwatches contain a calibrated accelerometer that samples, digitizes, and stores movement activity. When interfaced with a computer, a scoring algorithm provides estimates of various sleep parameters. The investigators will average data across each two-week assessment period to determine actigraphy-based WASO, Total Sleep Time (TST) and SE. Not all participants completed actigraphy procedures
Time Frame: Baseline to 8 week
Population: To be included in actigraphy analyses, actigraphy data must have overlapped with sleep diary data (same dates) for a minimum of 7 nights. Estimated means were used. This is an intention to treat analysis. All subjects who completed baseline were included in analysis. Estimated means were calculated from a linear mixed model and used for the analysis.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 74 | 74
minutes
  Baseline | 5.9 (0.1) | 5.9 (0.1)
  8 week: number analyzed (Participants) | 54 | 63
  8 week | 6.2 (0.2) | 6.2 (0.2)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Test type: Equivalence — alpha = .05; p > 0.05, Mixed Models Analysis — alpha =.05; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-.4 to .5]

7. Secondary Outcome: Objective Sleep Efficiency (SE)
Description: Objective SE using Wrist Actigraphy. The investigators will use Actiwatch (Respironics, Inc.) wristwatch style actigraphs for collecting objective sleep data. Actiwatches contain a calibrated accelerometer that samples, digitizes, and stores movement activity. When interfaced with a computer, a scoring algorithm provides estimates of various sleep parameters. SE is the percentage of time spent in bed sleeping, scored total sleep time divided by (interval duration minus total invalid time (sleep/wake)) of the given rest interval multiplied by 100.The investigators will average data across each two-week assessment period.
Time Frame: Baseline to 8 week
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percentage of time in bed where asleep
Arm/Group | Tele-Self CBTI | Health Education Control
Number analyzed (Participants) | 74 | 74
percentage of time in bed where asleep
  Baseline | 86.3 (0.4) | 86.3 (0.4)
  8 week: number analyzed (Participants) | 54 | 63
  8 week | 87.0 (0.6) | 85.4 (0.5)
Statistical Analysis 1: Comparison: Tele-Self CBTI vs Health Education Control; Test type: Equivalence — alpha = .05; p < 0.05, Mixed Models Analysis — alpha = .05; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.2 to 2.9]

ADVERSE EVENTS:
Time Frame: from randomization to 6 month assessment, approximately 6 months.
Description: Participants were queried at Baseline, 8 weeks and 6 months.
Arm/Group | Tele-Self CBTI | Health Education Control
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/90
Serious Adverse Events (participants affected / at risk) | 15/88 | 16/90
Other Adverse Events (participants affected / at risk) | 31/88 | 37/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-Self CBTI (N=88) | Health Education Control (N=90)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 3 (3) | 1 (1) — Infections and infestations
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 2 (2)
renal (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Surgical and medical procedures (Surgical and medical procedures) | 4 (4) | 6 (6)
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-Self CBTI (N=88) | Health Education Control (N=90)
Blood and Lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 2 (2)
General (General disorders) | 1 (1) | 7 (7) — 2 HEC were study related; 1 disappointment at group assignment and 1 delay at being paid
Infections and infestations (Infections and infestations) | 7 (8) | 9 (11)
Injury and procedural complications (Injury, poisoning and procedural complications) | 6 (8) | 5 (6) — 3 INT and 5 HEC events were study-related (skin irritation from wrist band)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Nervous system disorders (Nervous system disorders) | 0 (0) | 3 (3)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 5 (5)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 1 (1)
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Social circumstances (Social circumstances) | 4 (4) | 6 (6)
Surgical and medical procedures (Surgical and medical procedures) | 4 (4) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 1 (1)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) — bells palsy

LIMITATIONS AND CAVEATS:
Limitations of the study include not achieving equal contact time across conditions and having lower retention of active arm than control condition participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03727438/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT03727438/ICF_001.pdf